CLINICAL TRIAL: NCT04070755
Title: A 6-Week, Randomized Study to Evaluate the Potential of FMX-101, 4% And Vehicle to Induce a Photo Allergic Skin Reaction in Healthy Volunteers, Using a Controlled Photo Patch Test Design
Brief Title: Dermal Photo Allergic Skin Reaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX2016-09
Record Dates: First submitted 2019-08-08; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMX-101 (Experimental)
  Interventions: Drug: FMX-101

INTERVENTIONS:
Drug: FMX-101

SUMMARY:
A 6-Week, Randomized Study to Evaluate the Potential of FMX-101, 4% And Vehicle to Induce a Photo Allergic Skin Reaction in Healthy Volunteers, Using a Controlled Photo Patch Test Design

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female who were 18 years of age or older
* Had uniformly-colored skin on the lower thoracic area of the back which allowed discernment of erythema, and were Fitzpatrick Skin Types I, II or III

Exclusion Criteria:

* Had any visible skin disease at the application site which, in the opinion of the investigative personnel, would have interfered with the evaluation of the test site reaction
* Had damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles or other disfigurations of the test site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-12-18 (Actual)

PRIMARY OUTCOMES:
Assessment of photoallergic skin reactions (numerical equivalent scoring of erythema and edema) after periodic exposure to IP on irradiated and non-irradiated skin | 6 weeks